CLINICAL TRIAL: NCT00338637
Title: Measuring the Balance Improvement on Multiple Sclerosis Patients After a Short Training Period With an APOS (All Phase Of Step Cycle) Kit
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-06-4127-AA-CTIL
Record Dates: First submitted 2006-06-19; First posted 2006-06-20 (Estimated); Last update posted 2006-06-20 (Estimated); Status verified 2006-06

CONDITIONS: Multiple Sclerosis; Balance; Cerebelar Impairment
MeSH Terms: conditions — Multiple Sclerosis

INTERVENTIONS:
Device: APOS shoe kit

SUMMARY:
Randomised double blind study of two parallel groups,one of the groups trained with the full APOS kit (a shoe with an additional bio mechanical device)

The control group trained with the Apos shoe without the bio mechanical device. both groups will be checked at the beginning of the study, one month later and at the end of the study after two months. The tests include neurological test, functional test(FSST,up and go test and berg balance test) gate analysis and quality fo life (rays) test.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Multiple sclerosis Cerebellar impairment EDSS under 4.5 age 18-65 years signed informed consent form

Exclusion Criteria:

* pregnancy
* coronary event in last 6 month
* 30 days or less after acute attack
* steroidal treatment in the last 60 days
* alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-04; Study Completion 2006-10

PRIMARY OUTCOMES:
functional tests

SECONDARY OUTCOMES:
gait analysis

CONTACTS AND LOCATIONS:
Overall Officials: Anat Achiron, Prof., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel